CLINICAL TRIAL: NCT05154019
Title: Managing Minds at Work: A Feasibility Pilot Cluster Randomised Control Trial for Online Interactive Training for Managers (Managing Minds at Work)
Brief Title: Managing Minds at Work: A Feasibility Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Institute of Mental Health Nottingham (Other); University of Warwick (Other); Loughborough University (Other)
Responsible Party: Principal Investigator, Louise Thomson, Associate Professor, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 299-0621
Record Dates: First submitted 2021-11-25; First posted 2021-12-10 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Occupational Stress; Occupational Neurosis; Mental Health Wellness 1; Absence; Sickness Behavior
Keywords: stress; mental health; line manager
MeSH Terms: conditions — Occupational Stress; Illness Behavior; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Waiting list control. Control group receive the training 3 months after completing baseline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Line Managers from organisations in the intervention arm will complete a self-led online training course consisting of 5 modules, over a period of 5-6 weeks
  Interventions: Behavioral: Managing Minds at Work Online Training
- Waitlist Control (No Intervention): Line Managers from organisations in the intervention arm will receive no training. They will be given access to the online intervention at the end of a 3-month period.

INTERVENTIONS:
Behavioral: Managing Minds at Work Online Training — The intervention will be an online, interactive training course which will include evidence-based material, guidance, and practical exercises. The training will cover the following topics, presented as a series of independent, stand-alone modules:
  Module one: Looking after your own mental health Module two: Designing and managing work to promote mental well-being Module three: Management Competencies that Prevent Work-related Stress Module four: Developing a Psychologically Safe Workplace Module five: Having conversations about mental health at work Each module will be designed to take between 20 and 30 minutes to complete. Participants will be permitted by their employer to complete the training within their work time. The training is self-led, so each participant can progress through each module at their own pace and at a time that suits them.
  Arms: Intervention

SUMMARY:
This feasibility pilot cluster RCT aims to pilot and feasibility test an online training toolkit (Managing Minds at Work) for line managers to develop their knowledge and confidence in preventing work-related stress and promoting mental health at work. The setting is work organisations of different types and sectors across the Midlands region of the United Kingdom. Participants must have direct managerial or supervisor responsibilities for 3 or more staff members.

The intervention consists of five modules of online learning: Looking after your own Mental Health; Designing and managing work to promote mental well-being; Management competencies to prevent work-related stress; Developing a psychologically safe work environment; Having conversations about mental health at work. Each module includes some descriptive content, interactive elements and opportunities for reflections, and take between 20-30 minutes to complete.

Participating organisations will be allocated to either the intervention or control arm. A waiting list control will be used, with line managers in the control organisations starting the intervention 3-months after baseline.

Data will be collected through online surveys with the intervention group at baseline, immediately post-intervention (around 6 weeks post baseline), 3-months follow-up and 6-months follow-up. Control group will complete the online surveys at baseline and 3-months (as they start the intervention) and immediately after completing the intervention. As a feasibility pilot study, analysis will be focused on acceptability of the intervention, feasibility of recruitment, retention and data collection, and estimating parameters for a larger trial. The primary outcome measure is line managers' confidence to create a mentally healthy workplace. The secondary outcomes line manger mental health knowledge, line manager workplace mental health literacy, line manager self-rating of behaviour. In addition, the direct reports of line managers will be invited to participate to assess the feasibility of collecting the outcome data related to: employee well-being, employee rating of line manager behaviour, employee sickness absence, employee productivity.

A process evaluation will be conducted to assess intervention acceptability, usability, implementation and effectiveness. Qualitative data will be collected via module feedback forms and in-depth interviews with a sample of line managers from the intervention arm and stakeholders.

DETAILED DESCRIPTION:
Study Aim

The overall aim of this project is to develop, pilot and feasibility test a new online training course (Managing Minds at Work) for line managers which provides guidance on preventing work-related stress and promoting mental health at work. This study will aim to assess the feasibility of a full cluster Randomised Controlled Trial (RCT) to assess the effectiveness of the training on improving line managers' outcomes (confidence, knowledge, behaviour) and employee outcomes (well-being, perceptions of line manager behaviours, sickness absence). In order to assess the feasibility and the potential effectiveness of the intervention, the study will test:

Study Objectives

The specific objectives are to test:

1. The potential for uptake within small, medium and large organisations by identifying and monitoring the:

   1. Willingness of employers to register interest in participating in the trial and allow line managers to take part in the trial.
   2. Recruitment and retention rates of line managers in the trial.
   3. Recruitment and retention of managers' direct reports.
2. The perceived suitability and effectiveness of the MMW intervention for line manager training by determining the:

   1. Acceptability, usability, and utility of the training among line managers and stakeholders within the participating organisations.
   2. Potential for improving line managers' confidence (primary outcome), knowledge and behaviours (secondary outcomes) to inform the planning of a larger trial.
   3. Potential for improving direct report outcomes (well-being, absence, self-reported productivity) by assessing changes to inform the planning of a larger trial.
3. The data collection methods for primary and secondary outcome measures to:

   1. Inform key parameters for a larger trial relating to sample size and clustering.
   2. Explore barriers and facilitators to the intervention implementation and effectiveness.

      Outcome Measures:
      * line managers confidence to create a mentally healthy workplace (primary)
      * line manger mental health knowledge
      * line manager workplace mental health literacy
      * line manager self-rating of behaviour
      * employee well-being
      * employee rating of line manager behaviour
      * employee sickness absence (organisational records)
      * employee productivity (self-reported)

      Study Design

      Cluster RCT Design This feasibility pilot study is a multi-site, two-armed cluster randomised controlled trial taking place in work organisations of different sizes and sectors across the Midlands area. The organisations are the units of randomisation (the clusters), with data collected from individual line managers (the participants) and the employees who work under their managers (their direct reports) within those organisations. If large, multi-site organisations are recruited to the study, the investigators will consider the option of using an internal control group within that organisation if there is a low risk of contamination between the intervention arm and control arm within that large organisation. The data collection schedule for the study is summarised in Table 2 and 3 below.

      Data Collection in Intervention Arm In the intervention arm, line managers will be invited to complete the online training course over a maximum period of 6 weeks. A repeated measures design will be adopted, whereby participants in the intervention arm will complete online questionnaires to collect data at baseline, on completion of the training (6 weeks), at 3 months follow-up and at 6-months follow-up. Line managers' direct reports will also be invited to complete online questionnaires at baseline, 3-months follow-up and 6-months follow-up. Where available, data will also be collected from organisational records on the sickness absence levels of employees managed by the participating line managers. Details of the measures in the online surveys are in the Outcome Measure section.

      Data Collection in Control Arm The study will employ a waitlist control, with line managers in the organisations within the control arm receiving the intervention after three months. Line managers in the control arm of the study will complete online questionnaires at baseline, just before the start of the training (3 months after baseline), immediately after completing the training (4.5 months after baseline). Line managers' direct reports will also be invited to complete online questionnaires at baseline and 3-months follow-up. Where available, data will also be collected from organisational records on the sickness absence levels of employees managed by the participating line managers. Details of the measures in the online surveys are in the Outcome Measure section

      Process Evaluation A qualitative process evaluation will run alongside the pilot trial to explore the experience of the intervention with line managers and other stakeholders within participating organisations, and assess the acceptability, usability and utility of the intervention and identify barriers and facilitators to implementation. Semi-structured interviews will be used to collect the data to inform the process evaluation. In addition, and module feedback forms will be completed by line managers after each of the modules in the training course to allow more specific feedback including any changes in their managerial practice that participants are planning to make as a result of completing the module.

      Randomization and Blinding Organisations (clusters) will be randomly assigned (1:1) to either the intervention or waiting list control group using an online random sequence generator (https://www.random.org/sequences/ ). This allocation will be stratified to ensure a spread of different size of organisations within the intervention and control arms. Where the organisation is sufficiently large to have distinct departments/divisions/units with minimal risk of contamination between them, the investigators will look to randomly assign two of these different departments/divisions/units to either intervention or the waiting list control using the same approach.

      The research team and participants will not be blinded to the outcome of randomisation due to practical reasons (i.e. sending reminder emails to participating managers).

      Selection and Withdrawal Of Participants Organisations The study setting will be any organisation with line managers and employees within the Midlands area. Participating organisations will be recruited through the communication channels (Twitter, Newsletters, Website). Organisations that register their interest will be receive a follow-up phone call from the lead researcher to provide further information about the study (Information Sheet for Organisation).

      Participants Managers within the participating organisations will be approached to participate in the study through a poster/flyer about the study, which will be shared with them by the gatekeeper within the organisation. Line managers who express interest in taking part will be given information about the study and asked to provide written consent prior to participating in the study (individual-level).

      Participating managers will be asked to share details of the study with their direct reports (people who they directly manage) to invite them to also participate in an online survey at baseline and 3 month follow-up.

      For the process evaluation interview study, participants will be invited to take part in interviews after the 6-month follow-up. Interviews will take place with:
      * Line managers in the intervention arm
      * Stakeholders (e.g. HR managers, Well-being co-ordinators etc) in both the intervention and control arms For line managers, on completing individual-level study consent all participants will have been asked to consent to being contacted by a qualitative researcher to take part in an interview. Those who have consented will be contacted and asked if they want to participate in a follow-up interview, and if so will be sent a PIS and consent form by email. Interviews will be conducted face-to-face, by video call or by telephone. Interviews will be arranged at a mutually convenient time and location.

      For stakeholders, the gatekeeper for each participating organisation (intervention and control arms) will be asked to email an invitation to participate in an interview to all relevant stakeholders within their organisation e.g. HR managers, well-being managers, learning and development managers, trade union representatives.

      Process Evaluation Interviews Semi-structured interviews will take place with line managers and direct reports from the intervention arm, and with stakeholders from both the intervention and control arm. These semi-structured interviews will be conducted with a random selection of participants following the completion of the training programme, to achieve a maximum variance sample based on size of organisation, sector, and participant demographics.

      Principles of data saturation will be used to guide the final sample size, but as a guideline the investigators would expect there to be interviews with approximately 20 line managers, 10 direct report, and 1 to 2 stakeholders per participating organisation. All of interviews and analysis will be conducted by member of the research team (CB, BV and KN). Interviews will be guided by the Interview Schedules and recorded using an encrypted digital recorder where consent is given. Digital audio files will be transferred to the transcription service Dict8 for transcription using secure FTP. Transcriptions will be anonymised. Audio files will be destroyed after transcripts have been checked. Anonymised transcriptions will be analysed and stored on the secure University of Nottingham server.

      Interviews with line managers

      The interview schedule will cover the following research questions and topics:
      * Acceptability, usability and utility of the intervention
      * Changes the line manager has introduced since undertaking the training
      * Barriers and facilitators to the intervention implementation and effectiveness
      * Suggested improvements to the intervention

      Interviews with stakeholders

      The interview schedule will cover the following research questions and topics:
      * Barriers and facilitators to taking part in the study
      * Acceptability of the wait-list control condition (control arm only)
      * Acceptability, usability and utility of the intervention
      * Barriers and facilitators to the intervention implementation and effectiveness

      Organisational Sickness Absence Records The investigators will collect information from the organisations regarding the sickness absence records of those the participating line managers directly manage. Pre-intervention data will cover the 6-months prior to the intervention. Post-intervention data will cover the 6-months post-intervention. All organisational absence records will be anonymised at source.

      Analyses

      Statistical Analysis and Sample size Statistical analysis will be produce summary statistics to assess the parameters for a full trial. Missing outcome data will be imputed using multiple imputation. SPSS will be used for statistical analysis.

      As this is a pilot trial, no emphasis will be put on the p values for any inferential statistical tests conducted. The pilot data will provide information on the parameters needed for a realistic sample size calculation (mean, standard deviation and treatment effects of the primary outcome for the two arms) for a future RCT. A minimum of 8 clusters (randomised into two groups of four) will be sought in order to inform a future trial.

      Process evaluation As part of the process evaluation additional qualitative data collection regarding the acceptability, usability, implementation, and effectiveness of the intervention will be collected through interviews with line managers, direct reports and stakeholders. The data collected analysed using thematic analysis within a framework approach.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Employed
* Direct managerial or supervision responsibility for three or more staff.
* Has a work computer or mobile phone and email address with which to access the training and receive reminders
* Ability to provide informed consent

Exclusion Criteria:

* Not employed
* Employed but due to retire or be made redundant in the next 6 months
* Have undertaken work-based training on mental health at work within last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
change in line managers confidence to create a mentally healthy workplace from baseline to 6 weeks | Baseline to 6 weeks follow-up
  Self-report scale assessing Confidence to Create Mentally Healthy Workplace (Gayed et al, 2109; Gayed et al, 2018). 6 items measured on 1 to 5 scale. Minimum value 5 (lowest confidence), maximum value 30 (highest confidence). Higher score means a better outcome.
change in line managers confidence to create a mentally healthy workplace from baseline to 3 months | Baseline to 3 months follow-up
  Self-report scale assessing Confidence to Create Mentally Healthy Workplace (Gayed et al, 2109; Gayed et al, 2018). 6 items measured on 1 to 5 scale. Minimum value 5 (lowest confidence), maximum value 30 (highest confidence). Higher score means a better outcome
change in line managers confidence to create a mentally healthy workplace from baseline to 6 months | Baseline to 6 months follow-up
  Self-report scale assessing Confidence to Create Mentally Healthy Workplace (Gayed et al, 2109; Gayed et al, 2018). 6 items measured on 1 to 5 scale. Minimum value 5 (lowest confidence), maximum value 30 (highest confidence). Higher score means a better outcome

SECONDARY OUTCOMES:
change in line manger mental health knowledge from baseline to 6 weeks | Baseline to 6 weeks follow-up
  Self-report scale assessing mental health knowledge (Evans-Lacko et al 2010). 6 items measured on 1 to 5 scale. Minimum value 5 (lowest knowledge), maximum value 30 (highest knowledge). Higher score means a better outcome
change in line manger mental health knowledge from baseline to 3 months | Baseline to 3 months follow-up
  Self-report scale assessing mental health knowledge (Evans-Lacko et al 2010). 6 items measured on 1 to 5 scale. Minimum value 5 (lowest knowledge), maximum value 30 (highest knowledge). Higher score means a better outcome
change in line manger mental health knowledge from baseline to 6 months | Baseline to 6 months follow-up
  Self-report scale assessing mental health knowledge (Evans-Lacko et al 2010). 6 items measured on 1 to 5 scale. Minimum value 5 (lowest knowledge), maximum value 30 (highest knowledge). Higher score means a better outcome
change in line manager workplace mental health literacy from baseline to 6 weeks | Baseline to 6 weeks follow-up
  Self-report survey assessing workplace mental health literacy (Moll et al, 2017). 16 items rating knowledge on a 1-5 scale. Minimum value 16 (lowest knowledge), maximum value 80 (highest knowledge). Higher score means a better outcome.
change in line manager workplace mental health literacy from baseline to 3 months | Baseline to 3 months follow-up
  Self-report survey assessing workplace mental health literacy (Moll et al, 2017). 16 items rating knowledge on a 1-5 scale. Minimum value 16 (lowest knowledge), maximum value 80 (highest knowledge). Higher score means a better outcome.
change in line manager workplace mental health literacy from baseline to 6 months | Baseline to 6 months follow-up
  Self-report survey assessing workplace mental health literacy (Moll et al, 2017). 16 items rating knowledge on a 1-5 scale. Minimum value 16 (lowest knowledge), maximum value 80 (highest knowledge). Higher score means a better outcome.
change in line manager self-rating of behaviour from baseline to 6 weeks | Baseline to 6 weeks follow-up
  Self-report survey assessing line management competencies (Management Competency Indicator Tool - manger version, HSE, 2009). 66 items rating behaviour on 1-5 scale. Minimum value 66 (lowest competencies), maximum value 330 (highest competencies). Higher score means a better outcome.
change in line manager self-rating of behaviour from baseline to 3 months | Baseline to 3 months follow-up
  Self-report survey assessing line management competencies (Management Competency Indicator Tool - manager version, HSE, 2009). 66 items rating behaviour on 1-5 scale. Minimum value 66 (lowest competencies), maximum value 330 (highest competencies). Higher score means a better outcome
change in line manager self-rating of behaviour from baseline to 6 months | Baseline to 6 months follow-up
  Self-report survey assessing line management competencies (Management Competency Indicator Tool - manager version, HSE, 2009). 66 items rating behaviour on 1-5 scale. Minimum value 66 (lowest competencies), maximum value 330 (highest competencies). Higher score means a better outcome
change in employee well-being from baseline to 3 months | Baseline and 3 months follow-up
  Self-report survey assessing well-being (Warwick-Edinburgh Mental Well-being Scale , Tennant et al, 2007). 14-items with a 1-5 response scale, minimum value 14 (low well-being) and maximum value 70 (high well-being). Higher score means a better outcome
change in employee well-being from baseline to 6 months | Baseline and 6 months follow-up
  Self-report survey assessing well-being (Warwick-Edinburgh Mental Well-being Scale , Tennant et al, 2007). 14-items with a 1-5 response scale, minimum value 14 (low well-being) and maximum value 70 (high well-being). Higher score means a better outcome
change in employee rating of line manager behaviour from baseline to 3 months | Baseline and 3 months follow-up
  Self-report survey assessing line management competencies (Management Competency Indicator Tool - employee version, HSE, 2009). 31 items rating behaviour on 1-5 scale. Minimum value 31 (lowest competencies), maximum value 155 (highest competencies). Higher score means a better outcome.
change in employee rating of line manager behaviour from baseline to 6 months | Baseline and 6 months follow-up
  Self-report survey assessing line management competencies (Management Competency Indicator Tool - employee version, HSE, 2009). 31 items rating behaviour on 1-5 scale. Minimum value 31 (lowest competencies), maximum value 155 (highest competencies). Higher score means a better outcome.
change employee sickness absence baseline to 6 months | Baseline and 6 months follow-up
  organisational records of sickness absence for direct reports of participating line managers. Higher score means worse outcome
change in employee productivity from baseline to 3 months | Baseline and 3 months follow-up
  self-reported 1-item scale completed by employees, minimum score 1 (usual productivity) and maximum value 5 (low productivity). Higher score means worse outcome
change in employee productivity from baseline to 6 months | Baseline and 6 months follow-up
  self-reported 1-item scale completed by employees, minimum score 1 (usual productivity) and maximum value 5 (low productivity). Higher score means worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Louise Thomson, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hassard J, Blake H, Dulal-Arthur TM, Frost A, Bartle C, Yarker J, Munir F, Vaughan B, Daly G, Meyer C, Russell S, Thomson L. Web-Based Interactive Training for Managers (Managing Minds at Work) to Promote Mental Health at Work: Pilot Feasibility Cluster Randomized Controlled Trial. JMIR Ment Health. 2025 Sep 2;12:e76373. doi: 10.2196/76373. PMID 40896820
- [Derived] Thomson L, Hassard J, Frost A, Bartle C, Yarker J, Munir F, Kneller R, Marwaha S, Daly G, Russell S, Meyer C, Vaughan B, Newman K, Blake H. Digital Training Program for Line Managers (Managing Minds at Work): Protocol for a Feasibility Pilot Cluster Randomized Controlled Trial. JMIR Res Protoc. 2023 Oct 24;12:e48758. doi: 10.2196/48758. PMID 37874612